CLINICAL TRIAL: NCT02356952
Title: A Low Glycemic Index Mediterranean Diet in the Treatment of Metabolic Syndrome. A Randomized Controlled Trial.
Brief Title: Effect of a Low Glycemic Index on Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera Specializzata in Gastroenterologia Saverio de Bellis (Other)
Responsible Party: Principal Investigator, Alberto R Osella, MD, PhD, Azienda Ospedaliera Specializzata in Gastroenterologia Saverio de Bellis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Medidiet
Record Dates: First submitted 2015-01-20; First posted 2015-02-06 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Metabolic Syndrome X
Keywords: Metabolic Syndrome X; Low Glycemic Index Mediterranean Diet; Low Glycemic Index Diet; Randomized Clinical Trial
MeSH Terms: conditions — Metabolic Syndrome | interventions — Diet, Mediterranean

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Mediterranean Diet (Experimental): Randomized prescription with indication about type of foods that can be consumed frequently (green foods), sometimes (yellow foods) and never (red foods).
  Interventions: Behavioral: Mediterranean Diet
- Low Glycemic Index Diet (Experimental): Randomized prescription with indication about type of foods that can be consumed frequently (green foods), sometimes (yellow foods) and never (red foods).
  Interventions: Behavioral: Low Glycemic Index Diet
- Low Glycemic Index Mediterranean Diet (Experimental): Randomized prescription with indication about type of foods that can be consumed frequently (green foods), sometimes (yellow foods) and never (red foods).
  Interventions: Behavioral: Low Glycemic Index Mediterranean Diet

INTERVENTIONS:
Behavioral: Mediterranean Diet — A list of foods that may be consumed frequently (green foods), sometimes (yellow foods) and never (red foods).
  Arms: Mediterranean Diet
Behavioral: Low Glycemic Index Diet — A list of foods that may be consumed frequently (green foods), sometimes (yellow foods) and never (red foods).
  Arms: Low Glycemic Index Diet
Behavioral: Low Glycemic Index Mediterranean Diet — A list of foods that may be consumed frequently (green foods), sometimes (yellow foods) and never (red foods).
  Arms: Low Glycemic Index Mediterranean Diet

SUMMARY:
Metabolic Syndrome (MetS) is a cluster of multiple risk factors of metabolic origin associated with an increased risk of cardiovascular disease, type 2 diabetes mellitus and other diseases, including some cancers. There has been an increased interest of researchers in the relationship between MetS and diet and, specifically, Mediterranean diet would be beneficial for people with high risk of developing MetS or individuals with established MetS.

DETAILED DESCRIPTION:
Metabolic Syndrome (MetS) is a cluster of multiple risk factors of metabolic origin, associated with an increased risk of cardiovascular disease, type 2 diabetes mellitus and other diseases, including some cancers. The National Cholesterol Education Program's Adult Treatment Panel III (NCEP-ATP III) defines MetS the presence of at least three of five diagnostic criteria consisting in the measure of waist circumference, fasting glucose, systolic pressure and/or diastolic blood pressure, serum triglycerides and HDL cholesterol. The level of physical activity, smoking habits, low social class membership as well as low level of education and even a mild degree of chronic inflammation have been associated with an increased risk of MetS. Recently, there has been an increased interest of researchers in the relationship between MetS and diet, and more specifically Mediterranean Diet (MD). A problem of the contemporary MD is the quality of carbohydrates as the foods rich in carbohydrates consumed actually, such as white bread and some type of pasta, are produced with refined flour, at high glycemic index (GI) and load (GL). There are numerous studies showing that taking large amounts of high GI and GL foods is a risk factor for coronary heart disease and type 2 diabetes. To our knowledge there is no diet trial that compared the health effects of Mediterranean diets with different quality of carbohydrates. Objective of this study was to compare, in a randomized clinical trial, the effects of a simple MD, a Low Glycemic Index diet (LGID), and a Low Glycemic Index MD (LGIMD) on MetS, MetS components and other metabolic variables. For this reason, after a baseline examination, participants were randomly divided into three groups, each receiving a specific dietary intervention, and all the parameters measured at the first visit were examined again at months third and sixth.

ELIGIBILITY:
Inclusion Criteria:

* MetS, Subject enrolled in the MICOL study in 2005-2006

Exclusion Criteria:

* Insulin treatment, Not enrolled in the MICOL study

Ages: 30 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2014-09; Primary Completion 2015-06 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in MetS score at six months | 6 months

SECONDARY OUTCOMES:
Change from Baseline in Serum Cholesterol at six months | 6 months
Change from Baseline in Serum HDL Cholesterol at six months | 6 months
Change from Baseline in Serum Triglycerides at six months | 6 months
Change from Baseline in Serum ALT at six months | 6 months
Change from Baseline in Serum Fasting Glucose at six months | 6 months
Change from Baseline in Serum insulin at six months | 6 months
Change from Baseline in Serum glycated hemoglobin at six months | 6 months
Change from Baseline in Systolic blood pressure at six months | 6 months
Change from Baseline in Diastolic blood pressure at six months | 6 months
Height | Baseline
Change from Baseline in Body Weight at six months | 6 months
Change from Baseline in Bioimpedenziometry at six months | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Rubén Osella, MD, PhD, Principal Investigator — IRCCS "Saverio De Bellis"; Giovanni Misciagna, MD, PhD, Study Director — IRCCS "Saverio De Bellis"
Locations (1):
- Laboratory of Epidemiology and Biostatistics-IRCCS Saverio de Bellis, Castellana Grotte, BA, Italy

IPD SHARING:
Plan to Share IPD: Undecided